CLINICAL TRIAL: NCT05414630
Title: A Prospective, Single-arm Clinical Study of Envafolimab as Consolidation Therapy in Patients With Locally Advanced/Unresectable (Stage III) Non-Small Cell Lung Cancer That Has Not Progressed After Concurrent/Sequential Chemoradiotherapy
Brief Title: A Study of Envafolimab in Subjects With Stage III Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yue-Yin Pan, The Professor of Anhui Provincial Cancer Hospital, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-NSCLC-009
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Non-small Cell Lung Cancer Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — envafolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab (Experimental): Envafolimab: subcutaneous injection, 300mg, Q3W
  Interventions: Drug: Envafolimab

INTERVENTIONS:
Drug: Envafolimab — Envafolimab: 300 mg，D1，Q3W, until PD or intolerable toxicity. The duration of treatment with Envafolimab should not exceed 2 years.

SUMMARY:
This is a prospective, single arm, phase II study to evaluate the efficacy and safety of Envafolimab in subjects with locally advanced/unresectable (Stage III) non-small cell lung cancer that has not progressed after prior concurrent/sequential chemoradiotherapy.

DETAILED DESCRIPTION:
Trial design: This is a single-arm, open-label trial in patients with locally advanced/unresectable (stage III) NSCLC who did not have disease progression after concurrent/sequential chemoradiotherapy to evaluate the efficacy of Envafolimab as a consolidation treatment of the efficacy and safety.

Background:The PACIFIC and GEMSTONE-301 studies have shown the efficacy of immunization as consolidation therapy in stage III NSCLC.

Patients with stage III NSCLC who did not have disease progression after at least two cycles of concurrent/sequential chemoradiotherapy (including platinum) will receive Envafolimab (300mg, Q3W, subcutaneous injection) within 1-42 days after the end of chemoradiotherapy. The maximum duration of Envafolimab treatment is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years.
2. Have histologically confirmed locally advanced/unresectable stage III non-small cell lung cancer.
3. The first dose of Envafolimab will be administered within 1-42 days (including 42 days) after concurrent/sequential chemoradiotherapy is completed.
4. ECOG performance status 0-2.
5. Life expectancy ≥ 12 weeks.
6. Adequate organ function.
7. For female subjects of childbearing age, urine or serum pregnancy test shall be conducted before receiving the first study drug administration, and the result is negative.
8. The subject and the subject's sexual partner need to use a medically approved contraceptive measure during the study treatment period and within 6 months after the end of the study treatment period.
9. Willing to participate in this trial; fully understand and informed of this trial, and able to provide written informed consent form (ICF).

Exclusion Criteria:

1. Disease progression after concurrent/sequential chemoradiotherapy.
2. Has received a live vaccine within 28 days prior to the first dose of investigational product.
3. Major surgical procedure (as determined by investigators) within 28 days prior to the first dose of investigational product.
4. Known positive driver gene mutation, such as EGFR sensitive mutation, ALK gene translocation or ROS1 rearrangement.
5. Received any antibody/drug targeting T-cell coregulatory proteins (immune checkpoints), with a washout period of less than 28 days.
6. Known history of human immunodeficiency virus (HIV) infection and/or acquired immune deficiency syndrome.
7. Subjects at active phase of chronic hepatitis B or with active hepatitis C.
8. History of organ transplantation.
9. History of inflammatory bowel disease or active inflammatory bowel disease (for example Crohn's disease or ulcerative colitis).
10. Severe allergic reaction to other monoclonal antibodies.
11. Subjects with other conditions that in the investigator's opinion may influence subject's compliance or make subjects not suitable for participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival (PFS) | 24 months after the last subject participating in.
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the date of randomization to the first date of recorded progression or all-cause death, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months after the last subject participating in.
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Objective Response Rate (ORR) | 24 months after the last subject participating in.
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects.
Duration of Response (DOR) | 24 months after the last subject participating in.
  DoR (per RECIST 1.1) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
Percentage of Patients Alive at 24 Months (OS24) | 24 months after the last subject participating in.
  OS24 was defined as the percentage of patients who were alive at 24 months after randomization per the Kaplan-Meier estimate of OS at 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Cancer Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No